CLINICAL TRIAL: NCT02470572
Title: Evaluation of the Omnyx™ Integrated Digital Pathology System in the Primary Diagnosis of Surgical Pathology Specimens
Acronym: PrimeDx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Omnyx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CD-0010
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Primary Diagnosis of Surgical Pathology Specimens

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omnyx™ IDP system (Active Comparator): Omnyx™ IDP system for Whole Slide Images (WSI)
  Interventions: Other: Omnyx™ IDP system
- Conventional light microscope (Placebo Comparator): conventional light microscope
  Interventions: Other: Conventional light microscope

INTERVENTIONS:
Other: Omnyx™ IDP system — Omnyx™ IDP system for Whole Slide Images (WSI)
  Arms: Omnyx™ IDP system
Other: Conventional light microscope — Conventional light microscope
  Arms: Conventional light microscope

SUMMARY:
A multi-site, randomized-read order, retrospective, paired-design evaluation of the Omnyx™ Integrated Digital Pathology (IDP) system with de-identified and previously signed-out cases from all major organ systems. Pathologist will read and diagnose cases on a conventional light microscope and on the Omnyx™ IDP system for Whole Slide Images (WSI) with a randomized read order. College of American Pathologists (CAP) cancer protocol checklists will be used to capture diagnostic reporting.

Diagnoses rendered by site Reading Pathologists will be captured on CAP checklists and compared directly to the Ground Truth (GT) diagnosis for both modalities.

DETAILED DESCRIPTION:
Following the FDA issued guidance document, "Informed Consent for In Vitro Diagnostic Device Studies Using Leftover Human Specimens that are Not Individually Identifiable"- 2006, the specimens are surgical pathology samples from leftover human specimens from clinical cases, archived and previously signed-out across the majority of surgical pathology subspecialties

ELIGIBILITY:
Inclusion Criteria:

• All surgical pathology samples from pre-identified list provided by FDA

Exclusion Criteria:

* Gross evaluation only specimens (including hardware and specimens that do not require microscopic review for diagnosis)
* Immunofluorescence specimens
* Fluid-based specimens
* Intraoperative consultation specimens only (frozen preparation)
* Specimens from which a slide(s) fails quality control according to user manuals and training and issue(s) cannot be remediated at the time of procurement and over-labeling; this includes having too many labels such that slide damage or scanner failure is likely (as outlined in Omnyx user manuals).
* Specimens for which any slide (other than a blank) that should be in the case part cannot be located

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of surgical pathology | 1 Year
  Demonstrate the effectiveness of the Omnyx™ IDP system is non-inferior to the Diagnostic Reference Standard glass diagnosis in routine surgical pathology cases.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Montalto, PhD, Study Chair — Omnyx, LLC

REFERENCES:
- See also: Company Website — http://www.omnyx.com